#### **Thesis**

Submitted for Partial Fulfillment of Master Degree in Clinical and Chemical Pathology

#### By

#### Mary Zakaria Fayek

*M.B*, *B.Ch*.

Misr University for Science and Technology (MUST)

#### **Under Supervision of**

#### **Prof. Dr. Mohamed Ameen Mekawy**

Professor of Clinical and Chemical Pathology

Faculty of Medicine- Ain-Shams University

#### Dr. Rasha Abd El-Rahman El-Gamal

Lecturer of Clinical and Chemical Pathology

Faculty of Medicine- Ain-Shams University

#### Dr. Ayman Abd Elkader Mohamed

Lecturer of Obstetrics and Gynecology
Faculty of Medicine- Ain -Shams University

#### Results

**Table (3):** Characteristics of patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELLP (n=24) | TTP/HUS (n=13) | Control (n=20) | $F/\chi^2$ | DF | p-value |
|---|---|---|---|---|---|---|
| Age (years) | $29.5 \pm 5.6$ | $25.3 \pm 4.5$ | $26.0 \pm 4.6$ | 4.086 | 2, 54 | 0.022¶† |
| Parity | | | | 0.213 | 1 | 0.645§ |
| P0 | 6 (25.0%) | 2 (15.4%) | 5 925.0%) | | | |
| P1 | 5 (20.8%) | 7 (53.8%) | 5 (25.0%) | | | |
| P2 | 8 (33.3%) | 2 (15.4%) | 6 (30.0%) | | | |
| Р3 | 2 (8.3%) | 1 (7.7%) | 3 (15.0%) | | | |
| P4 | 2 (8.3%) | 1 (7.7%) | 1 (5.0%) | | | |
| P5 | 1 (4.2%) | 0 (0.0%) | 0 (0.0%) | | | |
| Previous abortions | | | | 1.319 | 1 | 0.251§ |
| Nil | 23 (95.8%) | 12 (92.3%) | 18 (90.0%) | | | |
| One | 1 (4.2%) | 1 (7.7%) | 1 (5.0%) | | | |
| Three | 0 (0.0%) | 0 (0.0%) | 1 (5.0%) | | | |
| Gestational age<br>(weeks) | $30.5 \pm 4.0$ ‡ | 29.8 ± 5.4‡ | $24.2 \pm 3.2$ | 14.597 | 2, 54 | <0.001¶ |

Data are mean  $\pm$  SD or number (%).

<sup>¶</sup>One-way analysis of variance (ANOVA).

<sup>§</sup>Chi-squared test for trend.

<sup>†</sup>No statistically significant difference among the three groups by the Schéffé post-hoc test.

<sup>‡</sup>P-value <0.05 versus Control group (Schéffé test).

**Table (4):** Hemoglobin level, hematocrit, and schistoctyte count in patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELLP<br>(n=24) | TTP/HUS (n=13) | Control (n=20) | F | DF | P-value |
|---|---|---|---|---|---|---|
| Hemoglobin (g/dl) | $10.5 \pm 1.6$ | 11.1 ± 1.9 | $11.4 \pm 1.2$ | 1.773 | 2, 54 | 0.180¶ |
| Hematocrit (%) | $32.3 \pm 5.7$ | $33.1 \pm 6.5$ | $34.9 \pm 3.3$ | 1.457 | 2, 54 | 0.242¶ |
| Schistocyte count (%) | 0.5~(0.0-1.2)† | 6.5 (0.8 – 17.6)†‡ | 0.0 (0.0 – 0.0) | 27.186 | 2 | <0.0001§ |

Data are mean  $\pm$  SD or median (interquartile range).

<sup>¶</sup>One-way analysis of variance (ANOVA).

<sup>§</sup>Kruskal-Wallis test.

<sup>†</sup>P-value <0.05 versus Control group (Conover test).

<sup>‡</sup>P-value <0.05 versus SPE/HELLP group (Conover test).



**Figure (4):** Box plot showing the total platelet count in patients with SPE/HELLP or TTP/HUS and normal controls. Box represents the range from the first to third quartile (interquartile range). Line inside the box represents the median (second quartile). Whiskers represent the range between the minimum and maximum values excluding outliers (rounded markers) and extreme observations (asterisks).

**Table (5):** Total platelet count, immature platelet count, and immature platelet fraction in patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELLP<br>(n=24) | TTP/HUS (n=13) | Control (n=20) | $\chi^2$ | D<br>F | P-value |
|---|---|---|---|---|---|---|
| Total platelet count (*1,000/mm³) | 121 (73 –<br>188.5)† | 53.0 (37.0 –<br>81.0)†‡ | 269.5 (235.0 –<br>337.0) | 35.333 | 2 | <0.0001 |
| Immature<br>platelet count<br>(*1,000/mm³)<br>A-IPC | 14.875 (11.781<br>- 22.151)† | 11.64 (6.410<br>- 21.238)† | 21.992 (16.945<br>- 25.431) | 10.362 | 2 | 0.006 |
| Immature platelet fraction (%)IPF-% | 13.0 (9.6 –<br>22.9)† | 19.5 (15.1 –<br>27.7)†‡ | 7.2 (6.2 – 11.1) | 18.897 | 2 | <0.0001 |

Data are median (interquartile range).

<sup>†</sup>P-value <0.05 versus Control group (Conover test).

<sup>‡</sup>P-value <0.05 versus SPE/HELLP group (Conover test).



**Figure (5):** Box plot showing the total platelet count in patients with SPE/HELLP or TTP/HUS and normal controls. Box represents the range from the first to third quartile (interquartile range). Line inside the box represents the median (second quartile). Whiskers represent the range between the minimum and maximum values excluding outliers (rounded markers).



**Figure (6):** Box plot showing the immature platelet count (IPC) in patients with SPE/HELLP or TTP/HUS and normal controls. Box represents the range from the first to third quartile (interquartile range). Line inside the box represents the median (second quartile). Whiskers represent the range between the minimum and maximum values excluding outliers (rounded markers).



**Figure (7):** Box plot showing the immature platelet fraction (IPF) in patients with SPE/HELLP or TTP/HUS and normal controls. Box represents the range from the first to third quartile (interquartile range). Line inside the box represents the median (second quartile). Whiskers represent the range between the minimum and maximum values.

**Table (6):** Prevalence of a low platelet count, high IPF, or high schistocyte count among patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELLP<br>(n=24) | TTP/HUS (n=13) | Control (n=20) | P-value¶ |
|---|---|---|---|---|
| Low total platelet count (<100,000/mm³) | 9 (37.5%) | 11 (84.6%) | 0 (0.0%) | <0.001 |
| High IPF (>11.2%) (Machin, 2010) | 14 (58.3%) | 10 (76.9%) | 5 (25.0%) | 0.008 |
| High schistocyte count (>0%) (Gina et al.,2011) | 14 (58.3%) | 11 (84.6%) | 0 (0.0%) | <0.001 |

Data are number (%).

<sup>¶</sup>Fisher's exact test.



**Figure (8):** Prevalence of a low platelet count, high IPF, or high schistocyte count among patients with SPE/HELLP or TTP/HUS and normal controls.

**Table (7):** Receiver-operating characteristic (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF or schistocyte count

Marker

| Index | IPF | Schistocyte count |
|---|---|---|
| Sample size | 37 | 37 |
| Positive group (TTP/HUS) | 13 (35.1%) | 13 (35.1%) |
| Negative group (SPE/HELLP) | 24 (64.9%) | 24 (64.9%) |
| Area under the ROC curve (AUC) | 0.692 (0.519 to 0.833) | 0.771 (0.603 to 0.893) |
| z statistic | 2.028 | 3.022 |
| P-value | 0.043¶ | 0.003¶ |
| Associated cut-off criterion | >15.9 % | >4.6 % |
| Sensitivity (%) | 76.92 (46.2 - 95.0) | 61.54 (31.6 - 86.1) |
| Specificity (%) | 66.67 (44.7 – 84.4) | 91.67 (73.0 – 99.0) |
| Positive predictive value (PPV, %) | 55.6 (30.8 - 78.5) | 80.0 (44.4 - 97.5) |
| Negative predictive value NPV, %) | 84.2 (60.4 - 96.6) | 81.5 (61.9 - 93.7) |

Diagnostic indices are presented as value (95% CI).

<sup>¶</sup>DeLong method.



**Figure (9):** Receiver-operating characteristic (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF.



**Figure (10):** Receiver-operating characteristic (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the schistocyte count.

**Table (8):** Comparison of the receiver-operating characteristic (ROC) curves for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF-% or schistocyte count

| | Marker | | | | |
|---|---|---|---|---|---|
| Index | IPF-% | Schistocyte count | Difference | Z | P-value¶ |
| Area under ROC | 0.692 (0.519 to | 0.771 (0.603 to | 0.079 (-0.171 to | 0.617 | 0.537 |
| (AUC) | 0.833) | 0.893) | 0.328) | | |

Diagnostic indices are presented as value (95% CI). ¶DeLong method.



**Figure (11):** Comparison of the receiver-operating characteristic (ROC) curves for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF or schistocyte count.

**Table (9):** Receiver-operating characteristic (ROC) curve analysis for discrimination between patients with TMA and normal controls using the IPF-% or schistocyte count

| Marker |
|--------|

| Index | IPF | Schistocyte count |
|---|---|---|
| Sample size | 57 | 57 |
| Positive group (TMA) | 37 (64.9%) | 37 (64.9%) |
| Negative group (normal controls) | 20 (35.1%) | 20 (35.1%) |
| Area under the ROC curve (AUC) | 0.820 (0.695 to 0.909) | 0.838 (0.716 to 0.922) |
| z statistic | 5.678 | 8.660 |
| P-value | <0.0001¶ | <0.0001¶ |
| Associated cut-off criterion | >8.1 % | >0 % |
| Sensitivity (%) | 86.49 (71.2 - 95.5) | 67.57 (50.2 - 82.0) |
| Specificity (%) | 65.00 (40.8 - 84.6) | 100.00 (83.2 - 100.0) |
| Positive predictive value (PPV, %) | 82.1 (66.5 - 92.5) | 100.0 (86.3 - 100.0) |
| Negative predictive value (NPV, %) | 72.2 (46.5 - 90.3) | 62.5 (43.7 - 78.9) |

Diagnostic indices are presented as value (95% CI).

¶DeLong method.



**Figure (12):** Receiver-operating characteristic (ROC) curve for discrimination between patients with TMA and normal controls using the IPF.



**Figure (13):** Receiver-operating characteristic (ROC) curve for discrimination between patients with TMA and normal controls using the schistocyte count.

**Table (10):** Comparison of the receiver-operating characteristic (ROC) curves for discrimination between patients with TMA and normal controls using the IPF or schistocyte count

| Index | IPF | Schistocyte count | Difference | Z | P-value¶ |
|---|---|---|---|---|---|
| Area under ROC (AUC) | 0.820 (0.695 to 0.909) | 0.838 (0.716 to 0.922) | 0.018 (-0.105<br>to 0.142) | 0.290 | 0.7722 |

Diagnostic indices are presented as value (95% CI).

<sup>¶</sup>DeLong method.



**Figure (14):** Comparison of the receiver-operating characteristic (ROC) curves for discrimination between patients with TMA and normal controls using the IPF or schistocyte count.

**Table (11):** Multivariable binary logistic regression analysis for the relation between the IPF-% and TTP/HUS with adjustment for the confounding effect of the gestational age

| Variable | Regression coefficient (B) | SE for B | Wald | P-value | Odds ratio<br>(OR) | 95% CI for<br>OR |
|---|---|---|---|---|---|---|
| IPF -% | 0.084 | 0.041 | 4.105 | 0.043 | 1.088 | 1.003 to<br>1.179 |
| Gestational age (weeks) | -0.064 | 0.087 | 0.539 | 0.463 | 0.939 | 0.792 to<br>1.112 |
| Constant | -0.271 | | | | | |

**Table (12):** Multivariable binary logistic regression analysis for the relation between the schistocyte count and TTP/HUS with adjustment for the confounding effect of the gestational age

| Variable | Regression coefficient (B) | SE for B | Wald | P-value | Odds ratio<br>(OR) | 95% CI for<br>OR |
|---|---|---|---|---|---|---|
| Scistocyte count (%) | 0.101 | 0.052 | 3.781 | 0.052 | 1.107 | 0.999 to<br>1.226 |
| Gestational age (weeks) | -0.052 | 0.088 | 0.355 | 0.551 | 0.949 | 0.799 to<br>1.127 |
| Constant | 0.420 | | | | | |

**Table (13):** Correlation between the IPF and schistocytes count in whole study population, patients with TMA, SPE/HELLP, or TTP/HUS, and normal controls

| | Correlation between IPF-% and schistocyte cou | | |
|---|---|---|---|
| Group | Number | Spearman rho (ρ) | P-value |

| All study population | 57 | 0.466 | 0.0003 |
|----------------------|----|--------|--------|
| TMA | 37 | 0.231 | 0.169 |
| SPE/HELLP | 24 | 0.190 | 0.375 |
| TTP/HUS | 13 | -0.058 | 0.851 |
| Control | 20 | 0.000 | - |



**Figure (15):** Scatter plot showing the correlation between the IPF and schistocyte count in the whole study population. Fitted lines represent local regression smoothing (LOESS) trend lines.



**Figure (16):** Scatter plot showing the correlation between the IPF and schistocyte count in patients with TMA or normal controls. Fitted lines represent local regression smoothing (LOESS) trend lines.



**Figure (17):** Scatter plot showing the correlation between the IPF and schistocyte count in patients with SPE/HELLP or TTP/HUS and normal controls. Fitted lines represent local regression smoothing (LOESS) trend lines.

The results of the present study are shown in tables (14-22) and figures (18-29).

**Let Comparison between patients with SPE/HELLP or TTP/HUS and normal controls regarding demographic features:** 

There was significant difference between the three studied groups regarding maternal age (P <0.05) and high significant difference between the three groups regarding gestational age (P <0.001). However, there was no significant difference between parity and previous abortions (P >0.05). On applying Schéffé post-hoc test revealed no statistically significant difference among the three groups regarding maternal age (P >0.05). However, regarding gestational age, the Schéffé test has revealed a significant difference between either patient group (SPE/HELLP or TTP/HUS) versus control group (P <0.05 for each) (Table 14).

**Table (14):** Characteristics of patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELL<br>P (n=24) | TTP/HUS (n=13) | Control (n=20) | F/χ <sup>2</sup> | DF | p-value |
|---|---|---|---|---|---|---|
| Age | $29.5 \pm 5.6$ | $25.3 \pm 4.5$ | $26.0 \pm 4.6$ | 4.086 | 2, 54 | 0.022¶† |
| (years) | | | | | | |
| Parity | | | | | | • |
| P0 | 6 (25.0%) | 2 (15.4%) | 5 (25.0%) | 0.213 | 1 | 0.645§ |
| P1 | 5 (20.8%) | 7 (53.8%) | 5 (25.0%) | | | |
| P2 | 8 (33.3%) | 2 (15.4%) | 6 (30.0%) | | | |
| Р3 | 2 (8.3%) | 1 (7.7%) | 3 (15.0%) | | | |
| P4 | 2 (8.3%) | 1 (7.7%) | 1 (5.0%) | | | |
| P5 | 1 (4.2%) | 0 (0.0%) | 0 (0.0%) | | | |
| Previous abortions | | | | | | |
| Nil | 23 (95.8%) | 12 (92.3%) | 18 (90.0%) | 1.319 | 1 | 0.251§ |
| One | 1 (4.2%) | 1 (7.7%) | 1 (5.0%) | | | |
| Three | 0 (0.0%) | 0 (0.0%) | 1 (5.0%) | | | |
| Gestation<br>al age<br>(weeks) | 30.5 ± 4.0‡ | 29.8 ± 5.4‡ | $24.2 \pm 3.2$ | 14.59<br>7 | 2,<br>54 | <0.001¶ |

Data are mean  $\pm$  SD or number (%).

§Chi-squared test for trend.

<sup>¶</sup>One-way analysis of variance (ANOVA).

†No statistically significant difference among the three groups by the Schéffé post-hoc test. ‡P-value <0.05 versus Control group (Schéffé test).

- **Let Comparison between patients with SPE/HELLP or TTP/HUS** and normal controls regarding to laboratory data:
- <u>1) Hemoglobin level:</u> There was no significant difference between the three groups regarding hemoglobin (P > 0.05) (Table 15).
- <u>2) Hematocrit level:</u> There was no significant difference between the three groups regarding hematocrit (P > 0.05) (Table 15).
- <u>3) Schistocytes count:</u> There was high significant difference between the three groups regarding schistocytes count (p < 0.001). Applying Conover test reveal; significant difference between SPE/HELLP and control, between TTP/HUS and control and between SPE/HELLP and TTP/HUS (**Table 15**), (**Figure 18**).

**Table (15):** Hemoglobin level, hematocrit, and schistocytes count in patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELLP<br>(n=24) | TTP/HUS (n=13) | Control (n=20) | F | DF | P-value |
|---|---|---|---|---|---|---|
| Hemoglobin (g/dl) | $10.5 \pm 1.6$ | 11.1 ± 1.9 | 11.4 ± 1.2 | 1.773 | 2, 54 | 0.180¶ |
| Hematocrit (%) | $32.3 \pm 5.7$ | $33.1 \pm 6.5$ | $34.9 \pm 3.3$ | 1.457 | 2, 54 | 0.242¶ |
| Schistocyte count (%) | 0.5<br>(0.0 – 1.2)† | 6.5 (0.8 –17.6)†‡ | 0.01 (0.0 – 0.03) | 27.186 | 2 | <0.0001§ |

Data are mean  $\pm$  SD or median (interquartile range).

§Kruskal-Wallis test.

†P-value <0.05 versus Control group (Conover test).

‡P-value <0.05 versus SPE/HELLP group (Conover test).

<sup>¶</sup>One-way analysis of variance (ANOVA).



**Figure (18):** Box plot showing the schistocyte count in patients with SPE/HELLP or TTP/HUS and normal controls.

- <u>4) Total platelet count:</u> There was high significant difference between the three groups regarding total platelet count (p < 0.001). Applying Conover test reveal; significant difference between SPE/HELLP and control, between TTP/HUS and control and between SPE/HELLP and TTP/HUS (**Table 16**), (**Figure 19**).
- <u>5) Immature platelet count A-IPC</u>: There was significant difference between the three groups regarding immature platelet count (p < 0.05). Applying Conover test reveal; significant difference between SPE/HELLP and control, between TTP/HUS and control (Table 16), (Figure 20).
- <u>6) Immature platelet fraction IPF-%:</u> There was high significant difference between the three groups regarding immature platelet fraction (p < 0.001). Applying Conover test reveal; significant difference between SPE/HELLP and control, between TTP/HUS and control and between SPE/HELLP and TTP/HUS (Table 16), (Figure 21).
- **Table (16):** Total platelet count, immature platelet count, and immature platelet fraction in patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELLP (n=24) | TTP/HUS (n=13) | Control (n=20) | χ² | DF | P-value |
|---|---|---|---|---|---|---|
| Total platelet count (*1,000/mm³) | 121 (73 –<br>188.5)† | 53.0 (37.0 –<br>81.0)†‡ | 269.5 (235.0<br>- 337.0) | 35.333 | 2 | <0.0001 |
| Absolute<br>Immature platelet<br>count (*1,000/mm³)<br>(A-IPC) | 14.875 (11.781 –<br>22.151)† | 11.64 (6.410 –<br>21.238)† | 21.992<br>(16.945 –<br>25.431) | 10.362 | 2 | 0.006 |
| Immature platelet<br>fraction (%)(IPF-<br>%) | 13.0 (9.6 –<br>22.9)† | 19.5 (15.1 –<br>27.7)†‡ | 7.2 (6.2 –<br>11.1) | 18.897 | 2 | <0.0001 |

Data are median (interquartile range).

†P-value <0.05 versus Control group (Conover test).

‡P-value <0.05 versus SPE/HELLP group (Conover test).



**Figure (19):** Box plot showing the total platelet count in patients with SPE/HELLP or TTP/HUS and normal controls.



**Figure (20):** Box plot showing the immature platelet count (IPC) in patients with SPE/HELLP or TTP/HUS and normal controls.



**Figure (21):** Box plot showing the immature platelet fraction (IPF) in patients with SPE/HELLP or TTP/HUS and normal controls.

- <u>Prevalence of a low platelet count (A-IPC):</u> There was high significant difference between the three groups regarding prevalence of a low platelet count (P < 0.001) (Table 17), (Figure 22).
- <u>Prevalence of high IPF-%</u>: There was significant difference between the three groups regarding prevalence of high IPF (P <0.05) (**Table 17**), (**Figure 22**).
- <u>Prevalence of high schistocyte count:</u> There was high significant difference between the three groups regarding prevalence of high schistocyte count (P <0.001) (Table 17), (Figure 22).

**Table (17):** Prevalence of a low platelet count, high IPF, or high schistocyte count among patients with SPE/HELLP or TTP/HUS and normal controls

| Variable | SPE/HELLP (n=24) | TTP/HUS (n=13) | Control (n=20) | P-value¶ |
|---|---|---|---|---|
| Low total platelet count (<100,000/mm <sup>3</sup> ) | 9 (37.5%) | 11 (84.6%) | 0 (0.0%) | <0.001 |
| High IPF-% (>11.2%) (Machin, 2010) | 14 (58.3%) | 10 (76.9%) | 5 (25.0%) | 0.008 |
| High schistocyte count (>1%) (Gina et al., 2011) | 14 (58.3%) | 11 (84.6%) | 0.01 (0.0%) | <0.001 |

Data are number (%).

¶Fisher's exact test.



**Figure (22):** Prevalence of a low platelet count, high IPF, or high schistocyte count among the studied groups.

#### **4** Receiver-operating characteristic (ROC) curve analysis

**Table (18):** Receiver-operating characteristic (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF or schistocytes count

| Index | Marker |
|-------|--------|

| | IPF | Schistocyte count |
|---|---|---|
| Positive group (TTP/HUS) | 13 (35.1%) | 13 (35.1%) |
| Negative group (SPE/HELLP) | 24 (64.9%) | 24 (64.9%) |
| Area under the ROC curve (AUC) | 0.692 (0.519 to 0.833) | 0.771 (0.603 to 0.893) |
| z statistic | 2.028 | 3.022 |
| P-value | 0.043¶ | 0.003¶ |
| Associated cut-off criterion | >15.9 % | >4.6 % |
| Sensitivity (%) | 76.92 (46.2 - 95.0) | 61.54 (31.6 - 86.1) |
| Specificity (%) | 66.67 (44.7 – 84.4) | 91.67 (73.0 – 99.0) |
| Positive predictive value (PPV, %) | 55.6 (30.8 - 78.5) | 80.0 (44.4 - 97.5) |
| Negative predictive value (NPV, %) | 84.2 (60.4 - 96.6) | 81.5 (61.9 - 93.7) |

Diagnostic indices are presented as value (95% CI).

• (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF-%: The optimal cutoff values for IPF-% for discrimination between patients with TTP/HUS or SPE/HELLP was >15.9 %. The sensitivity and specificity were 76.92% and 66.7%, respectively. The positive predictive value (PPV) and negative predictive value (NPV) were 55.6 % and 84.2%, respectively (AUC=0.692) (Table 18) (Figure 23).

<sup>¶</sup>DeLong method.



**Figure (23):** Receiver-operating characteristic (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF.

• (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the schistocyte count: The optimal cutoff values for schistocyte count for discrimination between patients with TTP/HUS or SPE/HELLP was >4.6 %. The sensitivity and specificity were 61.54 % and 91.67%, respectively. The positive predictive value (PPV) and negative predictive value (NPV) were 80% and 81.5%, respectively (AUC=0.771) (Table 19), (Figure 24).



**Figure (24):** Receiver-operating characteristic (ROC) curve analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the schistocyte count.

#### Comparison of the receiver-operating characteristic (ROC) curves:

Comparison of the receiver-operating characteristic (ROC) curves between IPF-% or schistocyte count revealed no significant difference between IPF-% and schistocyte count regarding discrimination between patients with TTP/HUS or SPE/HELLP (P-value >0.05) (**Table 19**), (**Figure 25**).

**Table (19):** Comparison of ROC curves for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF or schistocyte count

| Index | IPF | Schistocyte count | Difference | Z | P-value¶ |
|---|---|---|---|---|---|
| Area under<br>ROC (AUC) | 0.692 (0.519<br>to 0.833) | 0.771 (0.603 to 0.893) | 0.079 (-0.171 to 0.328) | 0.617 | 0.537 |

Diagnostic indices are presented as value (95% CI).

<sup>¶</sup>DeLong method.



**Figure (25):** Comparison of ROC curves for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF or schistocyte count.

**Table (20):** ROC curve analysis for discrimination between patients with TMA and normal controls using the IPF-%s or schistocyte count

| Index | IPF-% | Schistocyte count |
|---|---|---|
| Positive group (TMA) | 37 (64.9%) | 37 (64.9%) |
| Negative group (normal controls) | 20 (35.1%) | 20 (35.1%) |
| Area under the ROC curve (AUC) | 0.820 (0.695 to 0.909) | 0.838 (0.716 to 0.922) |
| z statistic | 5.678 | 8.660 |
| P-value | <0.0001¶ | <0.0001¶ |
| Associated cut-off criterion | >8.1 % | >0 % |
| Sensitivity (%) | 86.49<br>(71.2 - 95.5) | 67.57 (50.2 - 82.0) |
| Specificity (%) | 65.00<br>(40.8 - 84.6) | 100.00 (83.2 - 100.0) |
| Positive predictive value (PPV, %) | 82.1 (66.5 - 92.5) | 100.0 (86.3 - 100.0) |
| Negative predictive value (NPV, %) | 72.2 (46.5 - 90.3) | 62.5 (43.7 - 78.9) |

Diagnostic indices are presented as value (95% CI).

¶DeLong method.

• (ROC) curve analysis for discrimination between patients with TMA or control using the IPF-%: The optimal cutoff values for IPF-% for discrimination between patients with TMA or control was >8.1%. The sensitivity and specificity were 86.49% and 65%, respectively. The positive predictive value (PPV) and negative predictive value (NPV) were 82.1 % and 72.2%, respectively (Table 20), (Figure 26).



**Figure (26):** ROC curve for discrimination between patients with TMA and normal controls using the IPF.

(ROC) curve analysis for discrimination between patients with TMA or control using schistocyte count: The optimal cutoff values for schistocyte count for discrimination between patients with TMA and normal controls was >0 %. The sensitivity and specificity were 67.57 % and 100%, respectively. The PPV and NPV were 100 % and 62.5%, respectively (Table 20), (Figure 27).



**Figure (27):** ROC curve for discrimination between patients with TMA and normal controls using the schistocyte count.

#### • Comparison of the receiver-operating characteristic (ROC) curves:

Comparison of the receiver-operating characteristic (ROC) curves between IPF-% or schistocyte count for discrimination between patients with TMA and normal controls revealed no significant difference between IPF and schistocyte count regarding discrimination between patients with TMA and controls (P > 0.05) (Table 21), (Figure 28).

**Table (21):** ROC curves for discrimination between patients with TMA and normal controls using the IPF or schistocyte count

| Index | IPF-% | Schistocyte count | Difference | Z | P-value¶ |
|---|---|---|---|---|---|
| Area under<br>ROC (AUC) | 0.820 (0.695<br>to 0.909) | 0.838 (0.716 to 0.922) | 0.018 (-0.105<br>to 0.142) | 0.290 | 0.7722 |

Diagnostic indices are presented as value (95% CI).

¶DeLong method



**Figure (28):** ROC curves for discrimination between patients with TMA and normal controls using the IPF or schistocyte count.

# **4** Correlation between IPF and schistocytes count with different parameters

no significant correlation was found between the IPF-% and schistocytes count in patients with SPE/HELLP, or TTP/HUS, as well as the whole TMA study group (Figure 29), (Table 22).

**Table (22):** Correlation between the IPF-% and schistocytes count in whole study population, patients with TMA, SPE/HELLP, or TTP/HUS, and normal controls

| | Correlation between IPF % and schistocyte count | | |
|---|---|---|---|
| Group | Number Spearman rho (ρ) P-value | | |
| ТМА | 37 | 0.231 | 0.169 |

| SPE/HELLP | 24 | 0.190 | 0.375 |
|-----------|----|--------|-------|
| TTP/HUS | 13 | -0.058 | 0.851 |



**Figure (29):** Scatter plot showing the correlation between the IPF and schistocyte count in patients with SPE/HELLP or TTP/HUS.

# IPF-% and schistocytes counts in TTP/HUS and SPE/HELLP using multivariate analysis

Multivariable binary logistic regression analysis was used for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF-% and schistocyte count combined. Both IPF-% (odds ratio, 1.11; 95% CI, 1.010 to 1.220; p= 0.031) and schistocyte count (odds ratio, 1.113; 95% CI, 1.016 to 1.219; p= 0.022) were independent predictors for TTP/HUS.

**Table (23):** Multivariable binary logistic regression analysis for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF and schistocyte count combined

| Variable | Regression<br>coefficient<br>(B) | SE<br>for B | Wald | P-<br>value | Odds ratio<br>(OR) | 95% CI for OR |
|---|---|---|---|---|---|---|
| IPF (%) | 0.104 | 0.048 | 4.666 | 0.031 | 1.110 | 1.010 to 1.220 |
| Schistocyte count (%) | 0.107 | 0.046 | 5.283 | 0.022 | 1.113 | 1.016 to 1.219 |
| Constant | -3.251 | | | | | |

**Table (24):** Receiver-operating characteristic (ROC) curve derived from the multivariable binary logistic regression model for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF-% and schistocyte count combined

| %) |
|----|
| %) |

| Value |
|------------------------|
| 0.827 (0.667 to 0.931) |
| 4.385 |
| <0.0001 |
| 92.3 (64.0 - 99.8) |
| 62.5 (40.6 - 81.2) |
| 2.46 (1.4 - 4.2) |
| 0.12 (0.02 - 0.8) |
| 57.1 (34.0 - 78.2) |
| 93.7 (69.8 - 99.8) |

Diagnostic indices are presented as value (95% CI). ¶DeLong method.



**Figure (30):** Discrimination between patients with TTP/HUS or SPE/HELLP using IPF-% and schistocyte count combined.

Table 24 and Figure 30 shows the results of ROC curve analysis derived from the predicted probabilities as estimated from the multivariable binary logistic regression model for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF and schistocyte count combined.

**Table (25):** Comparison of the receiver-operating characteristic (ROC) curves for discrimination between patients with TTP/HUS or SPE/HELLP using the IPF, schistocyte count, or IPF and schistocyte count combined

| Marker | AUC | 95% CI |
|-------------------|-------|----------------|
| IPF-% | 0.692 | 0.519 to 0.833 |
| Schistocyte count | 0.771 | 0.603 to 0.893 |

IPF-% and schistocyte count combined

0.827

0.667 to 0.931

| Marker | Difference<br>between AUCs | 95% CI | Z statistic | p-value |
|---|---|---|---|---|
| IPF-% vs. Schistocyte count | 0.079 | -0.171 to 0.328 | 0.617 | 0.537 |
| IPF-% vs. IPF and Schistocyte count combined | 0.135 | -0.034 to 0.303 | 1.569 | 0.117 |
| Schistocyte count vs. IPF-% and schistocyte count combined | 0.056 | -0.085 to 0.197 | 0.780 | 0.435 |



Figure (31): Discrimination between patients with TTP/HUS or SPE/HELLP.

The model had good predictive value as evidenced by increased AUC of 0.827 (95% CI, 0.667 to 0.931). The estimated sensitivity was 92.3% (64.0% - 99.8%), specificity of 62.5% (40.6% - 81.2%), PPV of 57.1%

(34.0% - 78.2%), and NPV of 93.7% (69.8% - 99.8%). However, no statistically significant difference (P >0.05) was revealed on comparing the AUC value of ROC curve of the combined use of IPF-% and schistocyte counts to AUC values of ROC curves of either marker alone for discrimination between patients with TTP/HUS or SPE/HELLP (Table 25, Figure 31).